CLINICAL TRIAL: NCT06519383
Title: Comparative Evaluation Of Accuracy Of Implant Position Achieved With Static Computer Assisted Fully Guided Implant Placement (sCAIP) And Conventional Cast Based Partially Guided Implant Placement (cPGIP)
Brief Title: Comparison Of Implant Position Achieved With Fully Guided Versus Partially Guided Implant Placement
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Krishnadevaraya College of Dental Sciences & Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 02_D012_00047
Record Dates: First submitted 2024-07-19; First posted 2024-07-25 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Implant Placement

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Implant placement by static computer assisted implant placement(fully guided). (Experimental): The Digital Imaging and Communications in Medicine (DICOM) file from the CBCT examination and the Standard Tessellation Language (STL) file from the surface scan will be imported and merged in planning software .The virtual implant planning for all patients will be performed in 3shape software.Surgical guide with embedded sleeve will be designed and 3D printed using computer-aided design/computer-aided manufacturing (CAD/CAM) technology.Fit and stability of static CAD\CAM surgical guide for test group will be verified through window areas of guide on top of the teeth.A flapless implant placement protocol will be performed for all implants.
  Interventions: Procedure: guided implant surgery
- Implant placement by conventional cast based partially guided implant placement(partially guided). (Experimental): A conventional acrylic stent with radiopaque marker (barium sulphate) will be fabricated which will serve as radiographic template.A CBCT (cone beam computed tomography) examination will be performed with the patient wearing radiographic template.The DICOM file will be then imported in planning software. Virtual implant planning will be performed in 3 shape software.A surgical stent will be produced in a conventional laboratory manner. A flapless implant placement protocol will be performed.
  Interventions: Procedure: guided implant surgery

INTERVENTIONS:
Procedure: guided implant surgery — Surgical guide is fabricated and fitted onto the patient's arch and implant is placed with guide in place.

SUMMARY:
Globally implant therapy is currently accepted as a predictable, viable and successful option to replace missing teeth. Ample studies have shown excellent survival and clinical success rates of dental implants for various indications.The correct three-dimensional (3D) positioning of an implant is considered a prerequisite for an optimal outcome.Computer assisted implant surgery maybe beneficial in patients with limited bone and proximity to anatomic structures.Therefore, the aim of this randomized controlled clinical trial is to investigate the accuracy of implant position achieved with static CAIP(Computer Assisted Implant Placement) and to compare this with the accuracy of conventional cast based partially guided implant placement(cPGIP).

DETAILED DESCRIPTION:
Globally implant therapy is currently accepted as a predictable, viable and successful option to replace missing teeth.As a result, the focus in contemporary implant dentistry has shifted towards the optimization of treatment concepts with aesthetics and function as an important outcome parameter.In this respect, implant installation should be prosthetically -driven, at the same time taking into account anatomical limitations as well as restrictions in terms of bone availability. Apart from aesthetics, a correct implant position may reduce biological and technical complications, favourable esthetic and prosthetic outcome, long term stability of peri-implant tissues, optimal occlusal contacts and implant loading. One possible tool that may facilitate a more accurate implant positioning is guided implant surgery.Virtual implant planning facilitates desired inter implant distance and depth. A top down planning wherein digital images of the edentulous area and mock wax up of the prosthesis is superimposed, allows precise implant placement planning. This digital planning can be converted into a surgical/virtual guide via a 3D printer or a milling machine.Fully guided surgery is based on a surgical guide which will assist the clinician in every step of the surgery starting from the first drill to the implant placement through the use of guiding sleeves in the guide. A partially-guided protocol differs only in the final step: after guided preparation of the osteotomy, the guide is removed and the implant is installed free-handedly.Therefore, the aim of this randomized controlled clinical trial is to investigate the accuracy of implant position achieved with static CAIP(Computer Assisted Implant Placement) and to compare this with the accuracy of conventional cast based partially guided implant placement(cPGIP).

ELIGIBILITY:
Inclusion Criteria:

* Patients in need of replacement of missing teeth.
* Mouth opening at least 30 mm.
* Age>18 years.
* Limited vertical or horizontal dimension of the alveolar ridge.
* Unfavorable bone morphology necessitating correct implant position.
* When minimally invasive (e.g. flapless) surgery is intended.
* When immediate implant restoration is planned.

Exclusion Criteria:

* Heavy smokers (more than 10 cigarettes per day)
* Uncontrolled diabetes
* Metabolic bone disorders
* History of radiotherapy of the head and neck
* Recent chemotherapy
* Use of drugs influencing bone or soft tissue healing (e.g., high doses of antiresorptive medication, steroids or anti-inflammatory drugs)
* Pregnant and/or lactating women

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Accuracy of implant position | 2 weeks
  3D deviation of planned implant position to final implant position